CLINICAL TRIAL: NCT04548531
Title: Engaging Patients in Colon Cancer Screening Decisions During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director of Health Decision Sciences Center, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020P001579-2
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-05

CONDITIONS: Colon Cancer
Keywords: Shared Decision Making; Colon Cancer Screening; COVID-19
MeSH Terms: conditions — Colonic Neoplasms; COVID-19 | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Two-armed randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Patients will not be given any information on their assigned arm. Statistician will be blinded to the assignment when analyzing the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Arm (No Intervention): This arm will be a usual care arm. Patients may call to schedule a colonoscopy or other tests as desired.
- Shared Decision Making Arm (Experimental): This is the intervention arm. Patients will receive a shared decision making information sheet in the mail and will be able to receive decision coaching from study staff to support selection of an option if desired.
  Interventions: Behavioral: Shared Decision Making

INTERVENTIONS:
Behavioral: Shared Decision Making — The decision aid is a paper information sheet presenting the pros and cons of three screening options (colonoscopy, stool-based tests, and postponing cancer screening until next year).
  The decision coaching is a structured interview to help patients clarify their preference for screening test and to support them in implementation (whether scheduling colonoscopy, ordering stool test or seeking additional advice from specialist).
  Other Names: Decision aid; Decision coaching
  Arms: Shared Decision Making Arm

SUMMARY:
The goal of the study is to examine whether a shared decision making intervention improves decision making about colon cancer screening for patients who had their colonoscopy delayed or postponed due to the COVID pandemic. Eligible patients (n=800) will be randomly assigned to either the intervention or control arm. A subset will be surveyed about 6-8 weeks post intervention to measure shared decision making, their intention to follow through with screening, and their decisional conflict. Study staff will conduct medical chart review to track receipt of colon cancer screening within 6 months. The statistician will test whether patients in the intervention arm report more shared decision making, less decisional conflict, higher intention to follow through on screening and have higher screening rates compared to those in the control arm.

DETAILED DESCRIPTION:
The goal of the study is to examine whether a shared decision making intervention improves decision making about colon cancer screening for patients who had their colonoscopy delayed or postponed due to the COVID pandemic. Eligible patient (n=800) will randomly assigned to either the intervention or control arm. A subset will be surveyed about 6-8 weeks post intervention to determine the extent to which they report shared decision making, their intention to follow through with screening, and their decisional conflict. Study staff will also conduct medical chart review to track receipt of colon cancer screening within 6 months.

Intervention arm: In this arm, patients will get a shared decision making information sheet in the mail that describes three screening options: (1) schedule next available colonoscopy, (2) switch to a stool-based test, and (3) delay colonoscopy for a year. Study staff trained in decision coaching will follow up with patients to help them select an option and support implementation.

Control arm: This arm will be a usual care arm. The gastroenterology department department has schedulers calling patients and texting patients to schedule their procedure.

All 800 patients will be followed for their cancer screening outcomes, and a subset n=460 or 230 in each arm will be randomly selected to receive the survey.

Study staff who prepare the intervention mailing and the surveys will not be blinded to the study arm. The staff who enter the data from the paper surveys and who conduct chart review to collect screening will be blinded to the assignment. The statistician analyzing the results will also be blinded to the assignment.

The following hypotheses will be evaluated using an intention to treat approach, so patients will be analyzed based on their assigned arm.

Hypothesis 1: Compared to the control group, patients in intervention arm will report higher shared decision making (primary outcome).

Hypothesis 2: Compared to the control group, patients in the intervention arm will have (2a) stronger intention to follow through with colon cancer screening (whether colonoscopy, stool-based test or other approach) and (2b) will be more likely to have a screening test within 6 months.

Hypothesis 3: Compared to the control group, patients in the intervention arm will have less decisional conflict (SURE score).

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 45-75
* Had screening or surveillance colonoscopy delayed or cancelled from March-June 2020

Exclusion Criteria:

* Diagnostic colonoscopy
* High risk for colorectal cancer as indicated by 1 year follow up schedule
* Prior history of colon cancer
* Unable to read or write in English or Spanish
* Have already scheduled or completed a colonoscopy since restrictions were lifted

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes To promote research replicability, transparency and future use of the data, de-identified data sets of the patient survey data will be created and will be available, by request, to outside researchers.
  After the main manuscripts have been published, de-identified data sets will also be deposited in an open access service such as, ICPSR (https://www.icpsr.umich.edu/icpsrweb/). Before a dataset is made available for access, ICPSR completes a detailed review of all datasets to assess disclosure risk. If necessary, ICPSR modifies data to reduce disclosure risk or limits access to datasets for which modifying the data would substantially limit their utility or the risk of disclosure remains high. No information that contains identifiers or that could be used to link an individual to the data will be included in the de-identified data set.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Three months after the end of the funded grant period, the study materials and de-identified data will be available, by request, from the PI. Once data are placed on an open access service such as ICPSR they will be available indefinitely.
Access Criteria: The PI will share a de-identified data set with outside investigators at no cost, according to approved Partners and Massachusetts General Hospital policies for data sharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.
  On ICPSR, individuals must register and agree to ICPSR's Responsible Use statement prior to accessing datasets.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On June 1, 2020, the co-investigators from the gastroenterology department extracted a list of patients aged 45-75, with preferred language of English or Spanish, who had a screening or surveillance colonoscopy that was cancelled, who had a referral for a screening colonoscopy that had not been processed, or who should have been contacted by the GI department to schedule a screening colonoscopy but had not been due to COVID-19 restrictions.
Groups:
- Usual Care (Control) Arm: This arm will be a usual care arm. Patients may call to schedule a colonoscopy or other tests as desired.
- Shared Decision Making (Intervention) Arm: This is the intervention arm. Patients will receive a shared decision making information sheet in the mail and will be able to receive decision coaching from study staff to support selection of an option if desired.
  Shared Decision Making: The decision aid is a paper information sheet presenting the pros and cons of three screening options (colonoscopy, stool-based tests, and postponing cancer screening until next year).
  The decision coaching is a structured interview to help patients clarify their preference for screening test and to support them in implementation (whether scheduling colonoscopy, ordering stool test or seeking additional advice from specialist).
Period: Intervention Period
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm
Started | 400 | 400
Completed | 399 | 399
Not Completed | 1 | 1
Period: 8-week Follow-up Survey
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm
Started | 252 (A random subset (n=252) of the 399 patients in each arm were selected to be mailed a survey to assess the intervention about 8 weeks later.) | 252 (A random subset (n=252) of the 399 patients in each arm were selected to be mailed a survey to assess the intervention about 8 weeks later.)
Completed | 124 | 119
Not Completed | 128 | 133

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm | Total
Number analyzed (Participants) | 399 | 399 | 798
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8) | 61 (8) | 60 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 217 | 424
  Male | 192 | 182 | 374
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 46 | 90
  Not Hispanic or Latino | 296 | 293 | 589
  Unknown or Not Reported | 59 | 60 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 19 | 14 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 18 | 43
  White | 292 | 298 | 590
  More than one race | 8 | 8 | 16
  Unknown or Not Reported | 55 | 60 | 115
Region of Enrollment [Number; unit: participants]
  United States | 399 | 399 | 798

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making (SDM) Process Scale Score
Description: short patient reported scale asks patients about discussion of options, pros and cons of colonoscopy and discussion of patients' preferences. Total scores range from 0-4 with higher scores indicating higher shared decision making.
Time Frame: About 8 weeks after intervention
Population: This analytic sample was a subset of the initial 798 patients at baseline who completed a survey about 8-weeks after the start of the intervention.
Measure: Mean (Standard Deviation); unit: Score on a scale of 0-4
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm
Number analyzed (Participants) | 124 | 119
Score on a scale of 0-4 | 0.27 (0.67) | 0.95 (1.27)
Statistical Analysis 1: Comparison: Usual Care (Control) Arm vs Shared Decision Making (Intervention) Arm; Test type: Superiority; p < .001, t-test, 2 sided; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [0.41 to 0.94]

2. Secondary Outcome: No Decisional Conflict (Number With Score of 4 on SURE Scale)
Description: The 4-item version of the decisional conflict scale, total score ranges from 0-4 and is reported as top score or percentage who score 4 which indicates no decisional conflict.
Time Frame: About 8 weeks after intervention
Population: This analytic sample was a subset of the initial 798 patients at baseline who were sent a survey about 8-weeks after the start of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm
Number analyzed (Participants) | 124 | 119
Participants | 52 | 73
Statistical Analysis 1: Comparison: Usual Care (Control) Arm vs Shared Decision Making (Intervention) Arm; Test type: Superiority; p = 0.003, Chi-squared; Risk Difference (RD) = 21, 95% CI 2-sided [7 to 35]

3. Secondary Outcome: Patient's Preferred Approach to Screening
Description: One item will assess patients' preferred approach to screening (with responses of colonoscopy, stool card test, no screening, not sure). We report on the percent of patients who had a clear preference for screening with either a stool card test or colonoscopy and those without a clear preference who chose no screening or not sure.
Time Frame: About 8 weeks after intervention
Population: This analytic sample was a subset of the initial 798 patients at baseline who were sent a survey about 8-weeks after the start of the intervention. There were 4 participants missing in the usual care arm and 7 patients missing in the intervention arm due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm
Number analyzed (Participants) | 120 | 112
Participants
  Patients with a clear preference (stool card test or colonoscopy) | 78 | 76
  Patients without a clear preference (unsure or no screening) | 42 | 36
Statistical Analysis 1: Comparison: Usual Care (Control) Arm vs Shared Decision Making (Intervention) Arm; We tested for a clear preference for screening, if a patient chose a colonoscopy or a stool-based test vs. the other response options; Test type: Superiority; p = .75, Chi-squared; Risk Difference (RD) = 3, 95% CI 2-sided [-10 to 16]

4. Secondary Outcome: Number Reporting "Very Likely" to Follow Through With Screening
Description: One item will assess patients' intention to follow through with their preferred approach on a 5-point scale from Very Unlikely to Very Likely. We report on the percent of patients who selected "Very Likely" to follow through with screening.
Time Frame: About 8 weeks after intervention
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm
Number analyzed (Participants) | 120 | 112
Participants | 87 | 94
Statistical Analysis 1: Comparison: Usual Care (Control) Arm vs Shared Decision Making (Intervention) Arm; We categorized for likelihood to follow through with screening. We reported on results from patients who indicated 'Very Likely' on their response option vs. the other options (likely, unsure, unlikely, very unlikely); Test type: Superiority; p = 0.14, Chi-squared; Risk Difference (RD) = 11, 95% CI 2-sided [-3 to 26]

5. Secondary Outcome: Colon Cancer Screening Rate
Description: Percentage of patients who had completed colon cancer screening test
Time Frame: 6 months after randomization
Population: At 6 months post-intervention, we assessed whether or not the 798 patients completed a colon cancer screening test.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm
Number analyzed (Participants) | 399 | 399
Participants | 91 | 140
Statistical Analysis 1: Comparison: Usual Care (Control) Arm vs Shared Decision Making (Intervention) Arm; Assessed how many patients completed any colorectal cancer screening test within 6-months after randomization; Test type: Superiority; p < .001, Chi-squared; Risk Difference (RD) = 13, 95% CI 2-sided [6 to 18]

ADVERSE EVENTS:
Time Frame: Patients were followed for 6 months.
Arm/Group | Usual Care (Control) Arm | Shared Decision Making (Intervention) Arm
All-Cause Mortality (participants affected / at risk) | 0/400 | 0/400
Serious Adverse Events (participants affected / at risk) | 0/400 | 0/400
Other Adverse Events (participants affected / at risk) | 0/400 | 0/400

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04548531/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT04548531/SAP_001.pdf